CLINICAL TRIAL: NCT06013397
Title: Clinical Trial of Ketogenic Diet in the Treatment of Mitochondrial Encephalomyopathy With Lactic Acidosis and Stroke-like Episodes(MELAS)
Brief Title: Effectiveness of Ketogenic Diet in MELAS Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0366
Record Dates: First submitted 2023-05-11; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-04

CONDITIONS: MELAS Syndrome; Ketogenic Dieting
MeSH Terms: conditions — MELAS Syndrome | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- self pre-and post-control (Experimental): It is a self pre- and post-control, which compares the outcomes of the ketogenic diet with the status that did not receive ketogenic treatment
  Interventions: Dietary Supplement: Ketogenic diet

INTERVENTIONS:
Dietary Supplement: Ketogenic diet — Ketogenic diet (KD) is a high-fat, low-carbohydrate and moderate protein diet pattern, suitable for refractory epilepsy, glucose carrier protein 1 deficiency, pyruvate dehydrogenase deficiency, tumors and some genetic metabolic diseases. The ketogenic diet has been used to treat epilepsy for nearly 100 years, and its safety has been recognized by the medical community. In 2015, the ketogenic diet was included in the "Clinical Diagnosis and Treatment Guidelines - Epilepsy Volume" and became a commonly used treatment for refractory epilepsy.

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of ketogenic diet in patients with MELAS syndrome. The main questions it aims to answer are:

Clarify the curative effects of ketogenic diet in the treatment of MELAS disease.

Prevent the aggravation of MELAS disease, and improve the quality of life of patients.

Provide reliable evidence-based medical basis for the clinical application of ketogenic diet in the treatment of MELAS syndrome patients.

The clinical data of the participants treated with ketogenic diet will be collected, including the completion of ketogenic diet and clinical data at the start of treatment and after 1 month, 3 months, 6 months and 12 months

DETAILED DESCRIPTION:
Ketogenic diet initiation and follow-up:

1. Before starting ketogenic diet treatment, patients with abnormal indexes such as liver, kidney, lipid, humoral immunity, hematuria, routine biochemical, electrolyte, trace elements and bone metabolism should be excluded, energy and nutrients should be calculated according to their height and weight, and patients will be taught with ketogenic diet treatment education
2. Patients were initiated ketogenic diet after a short period of fasting (fasting no more than 48 hours). After treatment was initiated, 13 of the calculated target energy was given on the first day, 23 of the target energy was given on the second day, and the target amount was reached on the third day. Nutritionists made appropriate adjustments to the target energy according to the level of blood keto measured by patients
3. Weekly follow-up via telemedicine system or social media, outpatient follow-up at the initiation of ketogenic therapy and at 1 month, 3 months, 6 months, and 12 months respectively. Outpatient follow-up was done in a joint clinic with a dietitian and a neurologist to evaluate the effects and side effects of ketogenic therapy on a compliant diet and related clinical examinations

Clinical data collection:

1. Demographic information and Medical history collection Gender, age, education level age of onset, genetic test, drug use, past history, personal history, family history
2. Clinical symptom collection According to the Newcastle Mitochondrial Disease Adult Scale(NMDAS), including migraine headaches, seizures, stroke-like episodes and etc.
3. Biochemical indicators Blood glucose, keto, lactate and pyruvate monitoring, dietary status, dietary ratio changes, energy changes, weight changes
4. Cognitive function assessment Cognitive function was assessed using Fepsy software
5. Diagnostic Examination Cranial MRI, scalp EEG

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the diagnostic criteria of MELAS and have received MELAS standard therapy but are not satisfied with the therapeutic effect, and voluntarily underwent ketogenic therapy

Exclusion Criteria:

* Diseases with porphyria and disturbances in fatty acid transport and oxidation, severe electrolyte metabolism abnormalities, severe hemodynamic instability, acute respiratory infections, uncontrolled systemic infections, severe liver and renal failure, cholesterolemia (>300mgdl), abnormal coagulation, acute pancreatitis, eating disorders, ketogenic diet intolerance, significant weight loss, poor compliance

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2038-06-01 (Estimated); Study Completion 2038-06-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Clinical Symptom Score in 1 Year | Baseline, 1 month, 3 months, 6 months and 12 months
  According to the newcastle mitochondrial disease adult scale(NMDAS), including migraine headaches, seizures, stroke-like episodes and etc.
Change from Baseline Biochemical indicators in 1 Year | Baseline, 1 month, 3 months, 6 months and 12 months
  Blood glucose
Change from Baseline Biochemical indicators in 1 Year | Baseline, 1 month, 3 months, 6 months and 12 months
  keto, lactate and pyruvate monitoring
Hamilton Anxiety Scale (HAMA) | Baseline, 1 month, 3 months, 6 months and 12 months
  Change from Baseline Cognitive Function in 1 Year. Cognitive function was assessed using "Fepsy" software
Hamilton Depression Scale(HAMD | Baseline, 1 month, 3 months, 6 months and 12 months
  Change from Baseline Cognitive Function in 1 Year . Cognitive function was assessed using "Fepsy" software
Wechsler Intelligence Scale(WISC) | Baseline, 1 month, 3 months, 6 months and 12 months
  Change from Baseline Cognitive Function in 1 Year . Cognitive function was assessed using "Fepsy" software
Mini-mental State Examination(MMSE) | Baseline, 1 month, 3 months, 6 months and 12 months
  Change from Baseline Cognitive Function in 1 Year . Cognitive function was assessed using "Fepsy" software
Change from Baseline Diagnostic Examination in 1 Year | Baseline, 1 month, 3 months, 6 months and 12 months
  Cranial MRI（multimodal） Scalp EEG to evaluate posterior head α rhythm, discharge index, interictal epileptic discharges

SECONDARY OUTCOMES:
Demographic Information and Medical History Collection | Baseline
  Gender, age, education level age of onset, genetic test, drug use, past history, personal history, family history

CONTACTS AND LOCATIONS:
Overall Officials: Shuang Wang, doctor, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China